CLINICAL TRIAL: NCT05279495
Title: Double-Blind Study Determining the Efficacy of CannaXR in Decreasing UVA Premutagenic and Photoaging Markers
Acronym: CNXR-001D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MINO Labs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CNXR-001D
Record Dates: First submitted 2022-02-05; First posted 2022-03-15 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Photoaging

STUDY DESIGN:
Intervention Model Description: Study Design: Prospective, double-blind, vehicle-controlled pilot study
Masking Description: Subjects will receive sufficient CANNAXR cream (CANNAXR pods filled with CBD) and VEHICLE cream (cream with empty CANNAXR pods without CBD) in pump containers, marked right or left. Contents of pump containers unknown to subjects and investigators. All 20 subjects are treated with CANNAXR and Vehicle and the exposed to 3X their individual MED-UVA. The masking relates to which hip (right or left) of each individual receives which treatment, CANNAXR or Vehicle. Therefore there is masking of the treatments of all 20 subjects receiving both treatments, considered by clinicaltrial.gov a single arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Loaded CANNAXR (Other): In a double-blinded fashion, 250 mg CANNAXR cream and 250 mg VEHICLE cream will be randomized for application to a delineated 50 cm2 area of either the left or right, hip/buttocks skin twice daily for 2 weeks.
  In a double-blinded fashion, 250 mg CANNAXR cream and 250 mg VEHICLE cream will be randomized for application to a delineated 50 cm2 area of either the left or right, hip/buttocks skin twice daily for 2 weeks.
  Interventions: Device: In a double-blinded fashion, 250 mg CANNAXR cream; Device: Topical VEHICLE cream

INTERVENTIONS:
Device: In a double-blinded fashion, 250 mg CANNAXR cream — Determining the Efficacy of topically applied CANNAXR cream in Decreasing UVA Premutagenic and Photoaging markers 8-oxo-dG and the common deletion. 250 mg TOPICAL CBD CANNAXR Cream will be randomized for application to a delineated 50 cm2 area of either the left or right, hip/buttocks skin twice daily for 2 weeks
  Other Names: TOPICAL CBD CANNAXR Cream
Device: Topical VEHICLE cream — Determining the Efficacy of topically applied VEHICLE cream in Decreasing UVA Premutagenic and Photoaging markers 8-oxo-dG and the common deletion. 250 mg VEHICLE cream will be randomized for application to a delineated 50 cm2 area of either the left or right, hip/buttocks skin twice daily for 2 weeks

SUMMARY:
Ultraviolet light A (UVA) causes oxidization of guanine to mutagenic 8-Oxoguanine (8-OxoG) and the most frequent and best characterized mutation in mitochondrial DNA (mtDNA), a deletion of 4,977 base pairs, called the "common deletion", a marker of photoaging.

DETAILED DESCRIPTION:
Evaluations & Schedule:

Clinical phase:

The study of each subject will last 4-5 weeks, with 7 visits (Screening visit 1, Baseline visit 2, Follow up visit 3, Follow up visit 4, Follow up visit 5 and Follow up/Final Visit 6).

Screening Visit:

Subjects will read and be explained the informed consent. Subjects who agree to participate will sign the informed consent and a copy will be given to them. Exclusion/inclusion criteria will be reviewed.

Subjects will be informed that the left arm will be photographed at visits 1 and 3 and both hip/buttock areas at each visit. A urine pregnancy test will be done on baseline (Visit 1, day 0) and final visit 6.

Visit 2, Baseline (day 0):

Baseline visit will be done no more than 21 days after the screening visit and may be done on the same day as the screening visit. Each subject will be instructed not to change any of his/her photoprotection practices during the duration of the study, including time spent outdoors each weekday and weekend day, with special attention between the hours of 10 AM and 4PM, and sunscreen use and parts of their body where they apply it.

The subject's left volar forearm will be exposed to 10, 15, 20, 25, 30, and 35 J/cm2 doses of ultraviolet A light, through a UVA opaque fenestrated adhesive patch placed, 2 cm distally from antecubital fossa. Appropriate UVA opaque shields will be used to protect surrounding untreated areas.

In double-blinded fashion, subjects will receive sufficient CANNAXR (extended release) cream (CANNAXR pods filled with CBD) and VEHICLE cream (cream with empty CANNAXR pods without CBD) in pump containers, marked right or left, with detailed application instructions and a template for each cream to be applied to specified 50 cm2 areas of either the left and right, hip/buttock skin daily in the morning and evening for 2 weeks, starting the next morning.

Visit 3 (Day 1):

MED-A (minimal erythema dose for UVA) will be determined by evaluating skin exposed the prior day to the different UVA doses. MED-A will be defined as the dose that produced "just perceptible erythema".

Visit 4 (Day 14) Subjects will be asked about adverse events (predicted or unpredicted, local or systemic) since the last visit. Within the treated areas of the right and left hip/buttock, skin will be treated through fenestrated adhesive UVA-opaque patches as follows: Window #1- no UVA dose, and Window #2 - 3x the subjects UVA-MED (determined on Day 1).

Visit 5 (Day 15):

Subjects will be asked about adverse events (predicted or unpredicted, local or systemic) since the last visit. Local anesthesia (lidocaine 2% with epinephrine) will be injected and a 4mm punch biopsy will be performed of the skin of each hip/buttock within the templated Windows #1 and #2, as well as at a site 10 cm from the treated area of the left hip/buttock. One or two 5-0 sutures will be placed to appose the skin edges at each of the biopsied sites. Skin biopsy specimens will be divided in half and placed in labelled containers containing appropriate media for 8-oxo-dG (8-oxo deoxyguanosine), common deletion, histochemical and immunochemical studies. Specimens will be shipped to Dr. Adam Friedman for analyses.

Supplies and wound care instructions will be given.

Visit 6, Final (Day 22-30):

Subjects will be asked about adverse events (predicted or unpredicted, local or systemic) since the last visit and all sutures placed at Visit 5 will be removed. A urine pregnancy test will be done.

Notes:

1. If an erythematous response after UVA light exposure is symptomatic (burning and tenderness), subjects will be allowed to use twice a day hydrocortisone 1%, over the counter cream, to treat the area. We will provide the cream at the office.
2. Visit 3 has to occur 20-28 hours after baseline visit 2.
3. Visit 5 has to occur 20-28 hours after Visit 4.

ELIGIBILITY:
Population:

Inclusion criteria:

* Healthy subjects
* 22-65 years of age
* Fitzpatrick skin types II and III

Exclusion criteria:

* Pregnancy
* Personal history of skin cancer
* History of abnormal photosensitivity
* Tobacco smoker
* History or being exposed to other forms of radiation (other than sunlight)
* Using any drug/medication that might alter the response of skin to UVA irradiation
* Unable to undergo skin biopsies
* History of abnormal scarring
* History of exposure to the treated areas with external beam X-ray or non-solar UV light irradiation

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Title: Double-Blind Study to measure and compare the Mean Percent Reduction UVA induced premutagenic and photoaging markers 8-oxo-dG and the common deletion in 20 subjects treated with CANNAXR and Vehicle and exposed to 3X their individual MED-UVA | 2 weeks
  Determining the Efficacy of topically applied CANNAXR cream vs vehicle cream in decreasing UVA induced Premutagenic and Photoaging markers 8-oxo-dG and the common deletion in 20 subjects exposed to 3X their individual MED-UVA: Comparison of mean percent reduction in UVA induced 8-Oxo-DG and common deletion in CANNAXR and Vehicle treated skin and exposed to 3X MED-UVA

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical and Cosmetic Research, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruls WA, van Weelden H, van der Leun JC. Transmission of UV-radiation through human epidermal layers as a factor influencing the minimal erythema dose. Photochem Photobiol. 1984 Jan;39(1):63-7. doi: 10.1111/j.1751-1097.1984.tb03405.x. No abstract available. PMID 6701210
- [Background] Wondrak GT, Jacobson MK, Jacobson EL. Endogenous UVA-photosensitizers: mediators of skin photodamage and novel targets for skin photoprotection. Photochem Photobiol Sci. 2006 Feb;5(2):215-37. doi: 10.1039/b504573h. Epub 2005 Aug 19. PMID 16465308
- [Background] Zhang X, Rosenstein BS, Wang Y, Lebwohl M, Mitchell DM, Wei H. Induction of 8-oxo-7,8-dihydro-2'-deoxyguanosine by ultraviolet radiation in calf thymus DNA and HeLa cells. Photochem Photobiol. 1997 Jan;65(1):119-24. doi: 10.1111/j.1751-1097.1997.tb01886.x. PMID 9066291
- [Background] 4. Appendix A. HW Lim, H Honigsmann, and JLM Hawk In Photodermatology, 2007. Informa Healthcare USA, INC. 443-445.
- [Background] Yarborough A, Zhang YJ, Hsu TM, Santella RM. Immunoperoxidase detection of 8-hydroxydeoxyguanosine in aflatoxin B1-treated rat liver and human oral mucosal cells. Cancer Res. 1996 Feb 15;56(4):683-8. PMID 8630995
- [Background] Agar NS, Halliday GM, Barnetson RS, Ananthaswamy HN, Wheeler M, Jones AM. The basal layer in human squamous tumors harbors more UVA than UVB fingerprint mutations: a role for UVA in human skin carcinogenesis. Proc Natl Acad Sci U S A. 2004 Apr 6;101(14):4954-9. doi: 10.1073/pnas.0401141101. Epub 2004 Mar 23. PMID 15041750
- [Background] Berneburg M, Gattermann N, Stege H, Grewe M, Vogelsang K, Ruzicka T, Krutmann J. Chronically ultraviolet-exposed human skin shows a higher mutation frequency of mitochondrial DNA as compared to unexposed skin and the hematopoietic system. Photochem Photobiol. 1997 Aug;66(2):271-5. doi: 10.1111/j.1751-1097.1997.tb08654.x. PMID 9277148